CLINICAL TRIAL: NCT06442267
Title: A Three-arm Randomized Controlled Non-inferiority Pilot Study Comparing Anticoagulation Strategies Using Unfractionated Heparin, Argatroban and Low-molecular-weight Heparin for Extracorporeal Membrane Oxygenation Support
Brief Title: Comparing Anticoagulation Strategies Using UFH, Argatroban and LMWH for ECMO Support
Acronym: CASUAL-ECMO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Johannes Gratz, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1644/2022
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Insufficiency; Circulatory Failure; Thromboembolism; Bleeding
Keywords: ECMO; Anticoagulation; Thromboembolic Event; Bleeding; extracorporeal life support; anticoagulant; heparin
MeSH Terms: conditions — Respiratory Insufficiency; Shock; Thromboembolism; Hemorrhage | interventions — argatroban; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Enoxaparin group (Experimental): Anticoagulation for the duration of the study will be conducted using subcutaneous Enoxaparin
  Interventions: Drug: Enoxaparin Injectable Solution
- Argatroban group (Experimental): Anticoagulation for the duration of the study will be conducted using intravenous Argatroban.
  Interventions: Drug: Argatroban, 1 Mg/mL Intravenous Solution
- Unfractionated heparin group (Active Comparator): Anticoagulation for the duration of the study will be conducted using intravenous unfractionated heparin
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Enoxaparin Injectable Solution — Subcutaneous Enoxaparin will be dosed at 0.5 mg/kg twice daily
  Arms: Enoxaparin group
Drug: Argatroban, 1 Mg/mL Intravenous Solution — Intravenous Argatroban will be administered as a continuous infusion of 0.1-1 µg/kg/min with a target modified thrombin time measured using Hemoclot of 0,40 - 0,60 µg/mL.
  Arms: Argatroban group
Drug: Unfractionated heparin — Unfractionated heparin will be administered as a continuous infusion of 7.5-20 units/kg/h with a target Anti FXa calibrated for UFH of 0.3-0.5 u/mL.
  Arms: Unfractionated heparin group

SUMMARY:
A three-arm randomized controlled non-inferiority pilot study comparing anticoagulation strategies using unfractionated heparin, argatroban and enoxaparin for extracorporeal membrane oxygenation support conducted as an investigator-initiated, prospective, parallel group, open-label, active comparator controlled, single center, phase IV study to evaluate the non-inferiority of enoxaparin or argatroban for anticoagulation during ECMO therapy in comparison to the current standard, unfractionated heparin, as measured by the incidence of thromboembolic events during the duration of ECMO therapy

ELIGIBILITY:
Inclusion Criteria:

* either

  * require ECMO support or
  * have been started on ECMO therapy within the last 12 hours

Exclusion Criteria:

* Patients exhibiting contraindications to anticoagulation in general or any of the three investigated substances
* Patients who are pregnant
* Patients suffering from a clinically relevant pre-existing coagulopathy
* Patients, for whom screening, randomization and implementation of study protocol cannot be initiated within 12 hours after cannulation
* Patients receiving ongoing therapeutic systemic anticoagulation prior to ECMO implantation, or exhibiting an indication for therapeutic anticoagulation (e.g., pulmonary embolism)
* Patients whose total duration of ECMO support lasts less than 24 hours
* Patients with start of ECMO support during CPR (eCPR)
* Patients with passive decarboxylation, without an active pumping system
* Patients, who have been weaned off ECMO support within the last 30 days
* Patients with central ECMO cannulation and/or after cardiopulmonary bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of thromboembolic events during ECMO therapy | through duration of the ECMO run; an average of 14 days
  Clinically relevant thromboembolic events (Clinical suspicion; confirmation via imaging)
  * Pulmonary embolism, deep vein thrombosis
  * Intracardiac thrombosis
  * Arterial thromboembolism including myocardial and cerebral infarction
  * Deep vein thrombosis (detected during daily routine sonography)
  * Need to exchange ECMO circuit due to acute or incipient clotting

SECONDARY OUTCOMES:
Bleeding events | through duration of the ECMO run; an average of 14 days
  Incidence of bleeding events classified according to BARC Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Gratz, PD, MD, PhD, Principal Investigator — Medical Univeristy of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria